CLINICAL TRIAL: NCT06647173
Title: Integrating a Combination HIV Prevention Intervention Into a Widely-Used Geosocial App for Chinese MSM: Pilot Study
Brief Title: The Blued+ Combination HIV Prevention Pilot Study in China
Acronym: Blued+
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); BlueD China (Unknown)
Responsible Party: Principal Investigator, Aaron Siegler, Associate Professor, Emory University
Other Study IDs: IRB00116983; R01AI143875 (NIH)
Record Dates: First submitted 2024-10-16; First posted 2024-10-17 (Actual); Results first posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Pre-Exposure Prophylaxis
Keywords: HIV Prevention; HIV Testing; Condom use; MSM; Dating Mobile Application

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Blued App: A three-month run-in period with the standard of care followed by the Blued+ intervention with participants for 12 months.
  Interventions: Behavioral: Blued+ Service Platform

INTERVENTIONS:
Behavioral: Blued+ Service Platform — During the intervention period, participants received the enhanced version of the Blued app. The free HIV prevention services were integrated into the Blued app: health messaging, in-home HIV testing, linkage to care for those testing HIV positive, condoms, lubricants, in-app screening, and provision to PrEP.

SUMMARY:
The proposed research includes a longitudinal pilot study to assess the feasibility and acceptability of Blued+. This combination HIV prevention intervention will integrate a combination package of HIV prevention services into Blued, a gay dating App, for men who have sex with men (MSM) in China.

Despite high HIV incidence among MSM, HIV prevention interventions such as pre-exposure prophylaxis (PrEP) use remains low in China. If the HIV prevention intervention services provided through the Blued+ App prove feasible and acceptable, the pilot test will facilitate the design of a larger study of intervention efficacy.

The study population will be self-reported HIV-negative Blued users who are 18 years of age or greater, were assigned a male sex at birth, report having anal sex with a man in the last 6 months, eligible for PrEP according to China's consensus statement, and reside in metropolitan Beijing or Chengdu, China.

DETAILED DESCRIPTION:
The pilot study will be an interrupted time series cohort of 400 MSM. In two cities, a three-month baseline standard of care (SOC) period with measurement at 0 and 3 months will be followed by a 12-month intervention period with the measurement at 6, 9, 12, and 15 months.

During the intervention, enrolled study participants will take surveys every 3 months, as well as have free access to the enhanced version of the Blued App, Blued+, which additionally provides HIV prevention intervention services such as HIV health messages, PrEP drugs, at-home HIV self-testing kits, condoms, and lubricants for no costs. Participants interested in PrEP will be required to have additional PrEP initiation physical exam clinical visits, follow-up clinical visits, and dry blood spot collection lab visits for blood PrEP level measurements.

The total study period is 15 months (3 months control run-in period and 12 months intervention). Online surveys are provided over the study period, 2 for the enrollment and basement, and 4 follow-ups for every 3 months of the intervention; physical exam visits are required for participants who chose to initiate and refill PrEP; 1 dry blood spot collection visit is provided for participants who chose to measure blood PrEP level.

The participants will be recruited online through the Blued App.

ELIGIBILITY:
Inclusion Criteria:

* Registered Blued app user
* ≥18 years of age
* Male sex at birth
* Self-report anal sex with a man in the last 6 months
* HIV-negative or unknown HIV status
* Behaviorally eligible for PrEP per published China guidance
* Able to complete study instruments in Mandarin Chinese
* Resident of the metropolitan area of Beijing or Chengdu, China
* Eligible for PrEP based on China's consensus statement
* Additional Inclusion criteria apply for PrEP

Exclusion Criteria:

* Not a registered Blued app user
* <18 years of age
* Not male sex at birth
* Does not report anal sex with a man in the last 6 months
* Has previously tested positive for HIV
* Not eligible for PrEP per published China guidance
* Unable to complete study instruments in Mandarin Chinese
* Not a resident of the metropolitan area of Beijing or Chengdu, China
* Currently enrolled in another HIV prevention study
* Evidence of fraudulent participation, such as a duplicate IP address, multiple screening attempts, duplicate emails, etc.
* Additional Inclusion criteria apply for PrEP

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study population includes registered Blued users who self-report male sex at birth, are age 18 years or older, who report anal sex with a man in the past 6 months, behaviorally eligible for PrEP, and who do not report an HIV diagnosis. Eligible men will be residents of metropolitan areas of Beijing or Chengdu, China.
Sampling Method: Non-Probability Sample
Enrollment: 423 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2024-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Siegler, PhD, Principal Investigator — Emory University
Locations (1):
- BlueD, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang W, Ning K, Koh SHE, Mi G, Yu F, Liu Y, Stegmueller D, Powers KA, Baral S, Sullivan PS, Siegler AJ. Integrating a Combination HIV Prevention Intervention Into a Widely Used Geosocial App for Chinese Men Who Have Sex With Men: Protocol for a Single-Arm Pilot and Repeated Cross-Sectional Study. JMIR Res Protoc. 2025 Sep 29;14:e69536. doi: 10.2196/69536. PMID 41021915

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Blued App
Started | 423
Completed | 399
Not Completed | 24
Not completed — Lost to Follow-up | 24

BASELINE CHARACTERISTICS:
Arm/Group | Blued App
Number analyzed (Participants) | 423
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 423
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 423
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  China | 423

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Blued+ in China
Description: The intervention will be determined to be feasible if a minimum proportion of participants receive services for home HIV testing (benchmark ≥30%) and PrEP initiation (benchmark ≥20%) through Blued+
Time Frame: 12 months after intervention initiation, 15 months after first study interaction
Population: Participants retained at endline
Measure: Count of Participants; unit: Participants
Arm/Group | Blued App
Number analyzed (Participants) | 399
Participants
  Participants receiving PrEP through Blued+ | 193
  Participants receiving HIV testing through Blued+ | 316

2. Primary Outcome: System Usability Scale (SUS)
Description: Acceptability of Blued+ in China will be measured using the System Usability Scale (SUS). The SUS is a widely used scale that evaluates the usability of products and systems through a 10-item question set. The total range of a score on this scale is 0 to 100. This scale does not have any sub-scales. Higher scores on this scale represent higher levels of intervention usability, with 100 being the highest usability and 0 being the lowest usability. Information on this scale and how to calculate values is found in: Bangor, Aaron, Philip T. Kortum, and James T. Miller. "An empirical evaluation of the system usability scale." Intl. Journal of Human-Computer Interaction 24.6 (2008): 574-594.
  The intervention will be considered acceptable if it reaches a total SUS rating score of ≥ 71/100, which has been interpreted as being 'good' usability.
Time Frame: 12 months after intervention initiation, 15 months after first study interaction
Population: Participants completing all items in the SUS scale
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Blued App
Number analyzed (Participants) | 343
score on a scale | 73.4 (14.4)

ADVERSE EVENTS:
Time Frame: Data were collected throughout the 12-month pilot study period.
Description: Definitions do not differ from clinical trials.gov definitions.
Arm/Group | Blued App
All-Cause Mortality (participants affected / at risk) | 0/423
Serious Adverse Events (participants affected / at risk) | 0/423
Other Adverse Events (participants affected / at risk) | 0/423

LIMITATIONS AND CAVEATS:
This was a pilot study with a single arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-07-17): https://cdn.clinicaltrials.gov/large-docs/73/NCT06647173/Prot_SAP_ICF_000.pdf